CLINICAL TRIAL: NCT04153201
Title: Effect of Hydroxychloroquine on Thrombosis Prevention and Antiphospholipid Antibody Levels in Patients With Primary Antiphospholipid Syndrome: An Pilot Randomized Prospective Study.
Brief Title: Hydroxychloroquine for Thrombosis Prevention and Antiphospholipid Antibody Reduction in Primary Antiphospholipid Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Maria Tektonidou, Associate Professor of Rheumatology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SC668/10062016
Record Dates: First submitted 2019-10-21; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Antiphospholipid Syndrome
Keywords: antiphospholipid antibody titers; thrombosis prevention; hydroxychloroquine; antimalarials; antiphospholipid syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Hydroxychloroquine; Antimalarials

STUDY DESIGN:
Intervention Model Description: 1 intervention arm (Hydroxychloroquine plus standard care), 1 control arm (standard care) Patients randomized 1:1 using block size 2 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental): Patients with primary antiphospholipid syndrome started on hydroxychloroquine while continuing standard care (vitamin K antagonists or direct oral anticoagulants, and/or antiplatelet agents, depending on primary APS subgroup)
  Interventions: Drug: Hydroxychloroquine
- Standard care (No Intervention): Patients with primary antiphospholipid syndrome continuing standard care only (vitamin K antagonists or direct oral anticoagulants, and/or antiplatelet agents

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 200 mg daily for patients weighing < 60 kg, hydroxychloroquine 400 mg daily for patients weighing >= 60 kg
  Other Names: Antimalarials; Plaquenil
  Arms: Hydroxychloroquine

SUMMARY:
This is an interventional drug study designed as a pilot for a randomized clinical trial, aimed at assessing the effect of hydroxychloroquine on the incidence rate of thrombosis in patients with primary antiphospholipid syndrome as the main outcome, as well as the safety of hydroxychloroquine administration in this population. In addition, the effect of hydroxychloroquine on antiphospholipid antibody titers will be assessed.

DETAILED DESCRIPTION:
Patients with primary antiphospholipid syndrome (either thrombotic or obstetric) on regular follow-up at our outpatient rheumatology department and being treated with standard care (systemic anticoagulants and/or antiplatelet agents), are randomized to receive either hydroxychloroquine plus standard care, or standard care alone, on a 1:1 ratio using block size 2 randomization, after exclusion of patients with contraindications to hydroxychloroquine or prior hydroxychloroquine use within 12 months of consideration for enrollment. Patients are monitored clinically every 3 months and the development of thrombosis and/or adverse effects attributable to hydroxychloroquine is recorded. Antiphospholipid antibody titers (anti-cardiolipin immunoglobulin G (IgG)/Immunoglobulin M (IgM) and anti-beta2-glycoprotein I IgG/IgM isotypes) are measured semi-annually. Intention-to-treat survival analysis is applied for assessing the effect of hydroxychloroquine on the incidence of thrombosis. Longitudinal mixed linear models are applied for assessing the effect of hydroxychloroquine on longitudinal titers of antiphospholipid antibodies.

ELIGIBILITY:
Inclusion Criteria:

Adult patients diagnosed with primary antiphospholipid syndrome (PAPS) [updated Sapporo criteria: Miyakis et al, J Thromb Haemost. 2006 Feb;4(2):295-306. PubMed 16420554]

Exclusion Criteria:

1. ≥4 American College of Rheumatology (ACR) classification criteria for Systemic Lupus Erythematosus (SLE)
2. ACR classification criteria for other systemic autoimmune disorders
3. active malignancy
4. treatment with Hydroxychloroquine (HCQ) in the previous 12 months
5. history of serious adverse events or contraindication to HCQ including a history of HCQ allergy, HCQ eye toxicity, or glucose-6-phosphate dehydrogenase deficiency, uncontrolled seizure disorder, liver enzyme elevation >2-fold the upper normal limit, and creatinine clearance <30ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01-15; Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Incident acute thrombosis in the venous or arterial circulation | 3 years
  incident acute arterial thrombosis (myocardial infarction, stroke, transient ischemic attack, occlusion of the peripheral limb and neck, splanchnic, or retinal arteries) or venous thrombosis (pulmonary embolism, deep vein thrombosis, splanchnic vein thrombosis, retinal vein occlusion) confirmed by appropriate imaging studies (doppler ultrasonography, computed tomography pulmonary angiogram, conventional angiography, magnetic resonance angiography, ventilation/perfusion lung scintigraphy)

SECONDARY OUTCOMES:
Hydroxychloroquine-related safety outcomes | 3 years
  * Retinal toxicity by ocular examination, visual field testing and optical coherence tomography yearly and upon reporting visual symptoms
  * Toxic myopathy: new onset motor strength <=4/5, myalgia and creatine kinase elevation
  * Liver toxicity: liver enzyme elevations >3x of upper limit of normal (ULN), or serum total bilirubin >2x ULN, with no cholestasis
  * Metabolism disorders (hypoglycemia, weight decrease) by quarterly body weight and blood glucose testing
  * Bone marrow suppression: drop in hemoglobin to < 10 mg/dl, white blood cells < 3700/μL, platelets < 150,000/μL according to a hematologist
  * Cardiac complications (conduction defects, QT prolongation, cardiomyopathy) screened by interview, physical examination, and semi-annual electrocardiogram
  * Seizures screened by interview and confirmed by electrocardiogram
  * Gastrointestinal upset, allergic reactions, skin reactions by interview and physical exam
Anticoagulation treatment-related safety outcomes | 3 years
  * Major bleeding, defined as fatal bleeding, or symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a fall in hemoglobin level of 2 g/dL or more, or leading to transfusion of two or more units of whole blood or red cells.
  * Minor bleeding defined as clinically evident bleeding not fulfilling the definition of major bleeding
General safety outcomes | 3 years
  * Hospitalization for any cause
  * Death of any cause
  * APS-related death (based on death certificate records)

OTHER OUTCOMES:
Antiphospholipid antibody titer variation | 3 years
  Anticardiolipin IgG antibody titers, anti-cardiolipin IgM antibody titers, anti-beta2-glycoprotein I IgG antibody titers, antibeta2-glycoprotein I IgM antibody titers measured every 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Maria G Tektonidou, MD PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Laikon General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Following publication of results in a medical journal, we are considering sharing data on longitudinal apl titers, demographic information, time to first thrombotic event, adverse events with hydroxychloroquine.
  General data protection rule (GDPR) of the European Union special requirements may apply.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will become available 6 months following publication of results, and will remain accessible for 2 years
Access Criteria: Individual patient data will be provided to researchers in order to perform relevant meta-analyses, after review and approval of the meta-analysis protocol. Potential publications of our results with the same data should be cited if sharing our data results in new publications.